CLINICAL TRIAL: NCT06759844
Title: A Randomized Controlled Clinical Study for Validating the Effectiveness of a Mobile Health Management Program Aimed At Colorectal Cancer Survivors with Comorbid Chronic Conditions
Brief Title: Effectiveness of a Mobile Health Management Program for Colorectal Cancer Survivors with Chronic Conditions
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: National Cancer Center, Korea (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-2024-4
Record Dates: First submitted 2024-11-13; First posted 2025-01-06 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2024-09

CONDITIONS: Diabetes Mellitus; Colo-rectal Cancer; Hypertension; Dyslipidemia
MeSH Terms: conditions — Diabetes Mellitus; Colonic Neoplasms; Hypertension; Dyslipidemias

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial evaluating the effectiveness of a mobile health application in colorectal cancer survivors with chronic conditions. The study does not involve any drug, biological product, or combination product.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Educational Booklet (Active Comparator): Basic content on chronic disease management is provided. The content includes a basic booklet on managing chronic diseases without specific strategies. It covers topics like maintaining a positive mindset, managing stress, and exercising.
  Interventions: Behavioral: Educational Booklet
- Mobile Health Application (Experimental): Participants in this arm will use a mobile health application designed for colorectal cancer survivors with comorbid chronic conditions. The application provides daily educational content, goal-setting features, and self-monitoring tools to promote healthy behaviors. It includes modules on exercise, dietary management, and adherence to a personalized health plan. Participants will use the app daily for 3 months, with weekly progress evaluations and feedback provided through the application interface.
  Interventions: Behavioral: Mobile Health Application

INTERVENTIONS:
Behavioral: Educational Booklet — A printed booklet containing general information on chronic disease management provided to participants for reference without interactive or digital features
  Arms: Educational Booklet
Behavioral: Mobile Health Application — A mobile health application that facilitates self-management of chronic conditions through daily education, personalized goal setting, and lifestyle monitoring. The intervention aims to improve participants' health behaviors and clinical outcomes by promoting active engagement with their health.
  Arms: Mobile Health Application

SUMMARY:
The goal of this clinical trial is to evaluate if a mobile health management program can improve chronic disease management among colorectal cancer survivors with comorbid conditions such as hypertension, diabetes, and dyslipidemia. The main questions it aims to answer are:

Does the mobile health application improve clinical outcomes such as blood pressure, blood glucose levels, and lipid profiles? Does the application enhance participants' health behaviors and self-management capabilities? Researchers will compare the mobile health application group to the educational booklet group to see if the digital intervention leads to better health outcomes and adherence to lifestyle changes

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 19 years or older Colorectal cancer survivors (patients within 5 years of completion of curative treatments such as surgery, radiation therapy, or chemotherapy) who also have chronic conditions (hypertension, dyslipidemia, or diabetes)

Specific registration criteria:

Diabetes: Fasting blood sugar (FBS) ≥ 126 mg/dL or HbA1c ≥ 6.5% Dyslipidemia: Low-density lipoprotein cholesterol (LDL) ≥ 130 mg/dL Hypertension: Systolic blood pressure (SBP) ≥ 140 mmHg or Diastolic blood pressure (DBP) ≥ 90 mmHg Individuals who understand the purpose of this study and provide informed consent to participate Individuals who own and use a smartphone (able to use an ICT-based health management program)

Exclusion Criteria:

* Individuals who are unable to speak, listen, or read in Korean Individuals determined by a physician to be physically or mentally unfit (e.g., shortness of breath, severe depression) to participate in the study Individuals who are deemed unable to use the ICT-based program

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Fasting Blood Sugar | From enrollment to the end of treatment at 3months
  Check for decreased blood sugar levels
Hemoglobin A1c | From enrollment to the end of treatment at 3months
  check if the level has decreased
Total Cholesterol | From enrollment to the end of treatment at 3months
  Check if the level has decreased
LDL Cholesterol | From enrollment to the end of treatment at 3months
  Check if the level has decreased
Systolic and Diastolic Blood Pressure | From enrollment to the end of treatment at 3months
  Check if the level has decreased
Body Weight | From enrollment to the end of treatment at 3months
  Check if the level has decreased
Body Mass Index | From enrollment to the end of treatment at 3months
  Check if the level has decreased
Physical Activity Levels | From enrollment to the end of treatment at 3months
  Check if the level has decreased

SECONDARY OUTCOMES:
Improvement in Health Management Capability | From enrollment to the end of treatment at 3months
  Differences in Questionnaire of Self-Assessment Tool
Increase in Health Behavior Patterns | From enrollment to the end of treatment at 3months
  Differences in Questionnaire of Health Behavior and Practice Index
Emotional and Subjective Health Status | From enrollment to the end of treatment at 3months
  Differences in Questionnaire of Patient Health Questionnaire-9

CONTACTS AND LOCATIONS:
Locations (1):
- SNU-SMG Boramae Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yun YH, Kang E, Cho YM, Park SM, Kim YJ, Lee HY, Kim KH, Lee K, Koo HY, Kim S, Rhee Y, Lee J, Min JH, Sim JA. Efficacy of an Electronic Health Management Program for Patients With Cardiovascular Risk: Randomized Controlled Trial. J Med Internet Res. 2020 Jan 22;22(1):e15057. doi: 10.2196/15057. PMID 32012053
- [Background] Shin S, Wook Shin D, Young Cho I, Jeong SM, Jung H. Status of dyslipidemia management and statin undertreatment in Korean cancer survivors: A Korean National Health and Nutrition Examination Survey study. Eur J Prev Cardiol. 2021 Jul 23;28(8):864-872. doi: 10.1177/2047487320905722. Epub 2020 Feb 23. PMID 34298552
- [Background] Shen Y, Wang C, Ren Y, Ye J. A comprehensive look at the role of hyperlipidemia in promoting colorectal cancer liver metastasis. J Cancer. 2018 Jul 30;9(16):2981-2986. doi: 10.7150/jca.25640. eCollection 2018. PMID 30123367
- [Background] Mills KT, Bellows CF, Hoffman AE, Kelly TN, Gagliardi G. Diabetes mellitus and colorectal cancer prognosis: a meta-analysis. Dis Colon Rectum. 2013 Nov;56(11):1304-19. doi: 10.1097/DCR.0b013e3182a479f9. PMID 24105007
- [Background] Park HC, Shin A, Kim BW, Jung KW, Won YJ, Oh JH, Jeong SY, Yu CS, Lee BH. Data on the characteristics and the survival of korean patients with colorectal cancer from the Korea central cancer registry. Ann Coloproctol. 2013 Aug;29(4):144-9. doi: 10.3393/ac.2013.29.4.144. Epub 2013 Aug 29. PMID 24032114
- [Background] Park HC, Jung KW, Kim BW, Shin A, Won YJ, Oh JH, Jeong SY, Yu CS, Lee BH. Characteristics and survival of korean anal cancer from the Korea central cancer registry data. Ann Coloproctol. 2013 Oct;29(5):182-5. doi: 10.3393/ac.2013.29.5.182. Epub 2013 Oct 31. PMID 24278855